CLINICAL TRIAL: NCT01537081
Title: Randomized, Double-Blind, Double Dummy, Placebo-Controlled Study of the Safety and Efficacy Mucinex (2400 mg/d) and Immediate-Release Guaifenesin (800 mg/d) in the Treatment of Symptoms of Acute Upper Respiratory Tract Infections For 7 Days
Brief Title: Safety and Efficacy of Mucinex and IR Guaifenesin the Treatment of Symptoms of Acute Upper Respiratory Tract Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-MUC-04
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2013-09-12 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-10

CONDITIONS: Acute Upper Respiratory Tract Infection
MeSH Terms: interventions — Acetylcysteine; Guaifenesin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mucinex 2400 mg/day (Experimental): The study is designed to meet regulatory requirement outside the US. The dosing regimen and assessments timepoints were dictated by IR GGE and do not match approved Mucinex labeling. Participants were instructed to take 2 Mucinex 600 mg tablets and 1 placebo tablet matching the 200 mg IR guaifenesin tablet by mouth, every 12 hours for 7 days. To ensure complete blinding, on Hours 6 and 18, this treatment group took 2 matching Mucinex placebo tablets combined with 1 IR guaifenesin placebo tablet.
  Interventions: Drug: Mucinex; Drug: Placebo
- Immediate-release Guaifenesin 800 mg/Day (Active Comparator): The dosing regimen and assessments timepoints were dictated by immediate-release guaifenesin (IR GGE). Participants were instructed to take 1 immediate-release guaifenesin (IR GGE) 200 mg tablet and 2 matching Mucinex placebo tablets by mouth, every 6 hours for 7 days.
  Interventions: Drug: Immediate-release Guaifenesin; Drug: Placebo
- Placebo (Placebo Comparator): Double dummy technique was employed requiring a large number of tablets and water to be consumed. Participants were instructed to take 2 matching Mucinex placebo tablets combined with 1 matching IR guaifenesin placebo tablet by mouth, every 6 hours for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mucinex — Mucinex combines immediate-release (IR) and modified-release guaifenesin in a bilayer tablet. Each tablet was 600 mg of guaifenesin and taken by mouth with a full glass of water.
  Other Names: Mucinex®; guaifenesin
  Arms: Mucinex 2400 mg/day
Drug: Immediate-release Guaifenesin — Each tablet was 200 mg of immediate-release (IR) guaifenesin and taken by mouth with a full glass of water.
  Other Names: IR guaifenesin; IR GGE
  Arms: Immediate-release Guaifenesin 800 mg/Day
Drug: Placebo — Placebo tablets in two formulations to match either Mucinex or IR guaifenesin taken by mouth with a full glass of water

SUMMARY:
The study is designed to meet regulatory requirement outside the US. The dosing regimen and assessments timepoints were dictated by immediate release (IR) guaifenesin (GGE) and do not match approved Mucinex labeling in the U.S. The purpose of this study is to determine whether Mucinex is effective and non-inferior as compared to placebo and immediate release guaifenesin in the treatment of symptoms of acute upper respiratory infections. This design was required based on EU regulatory guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Has developed cold symptoms within 3 days prior to dosing on Day 1.

Exclusion Criteria:

1. Chronic illnesses.
2. Febrile illness > 101 F within 7 days prior to Day 1,
3. Pregnant.
4. Known current malignancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2810 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Reckitt Benckiser Study Site, Hoover, Alabama
  - Reckitt Benckiser Study Site, Bell Gardens, California
  - Reckitt Benckiser Study Site, Harbor City, California
  - Reckitt Benckiser Study Site, Long Beach, California
  - Reckitt Benckiser Study Site, Sacramento, California
  - Reckitt Benckiser Study Site, San Francisco, California
  - Reckitt Benckiser Study Site, San Luis Obispo, California
  - Reckitt Benckiser Study Site, Colorado Springs, Colorado
  - Reckitt Benckiser Study Site, Denver, Colorado
  - Reckitt Benckiser Study Site, Daytona Beach, Florida
  - Reckitt Benckiser Study Site, Edgewater, Florida
  - Reckitt Benckiser Study Site, Largo, Florida
  - Reckitt Benckiser Study Site, Chicago, Illinois
  - Reckitt Benckiser Study Site, Normal, Illinois
  - Reckitt Benckiser Study Site, Wichita, Kansas
  - Reckitt Benckiser Study Site, Lexington, Kentucky
  - Reckitt Benckiser Study Site, Metairie, Louisiana
  - Reckitt Benckiser Study Site, New Orleans, Louisiana
  - Reckitt Benckiser Study Site, Brighton, Massachusetts
  - Reckitt Benckiser Study Site, Fall River, Massachusetts
  - Reckitt Benckiser Study Site, Bellevue, Nebraska
  - Reckitt Benckiser Study Site, Omaha, Nebraska
  - Reckitt Benckiser Study Site, Las Vegas, Nevada
  - Reckitt Benckiser Study Site, Rochester, New York
  - Reckitt Benckiser Study Site, Raleigh, North Carolina
  - Reckitt Benckiser Study Site, Cincinnati, Ohio
  - Reckitt Benckiser Study Site, Middleburg Heights, Ohio
  - Reckitt Benckiser Study Site, Warwick, Rhode Island
  - Reckitt Benckiser Study Site, Greer, South Carolina
  - Reckitt Benckiser Study Site, Dakota Dunes, South Dakota
  - Reckitt Benckiser Study Site, Franklin, Tennessee
  - Reckitt Benckiser Study Site, Jackson, Tennessee
  - Reckitt Benckiser Study Site, New Tazewell, Tennessee
  - Reckitt Benckiser Study Site, Smyrna, Tennessee
  - Reckitt Benckiser Study Site, Austin, Texas
  - Reckitt Benckiser Study Site, Carrollton, Texas
  - Reckitt Benckiser Study Site, Forth Worth, Texas
  - Reckitt Benckiser Study Site, San Angelo, Texas
  - Reckitt Benckiser Study Site, Tomball, Texas
  - Reckitt Benckiser Study Site, Salt Lake City, Utah
  - Reckitt Benckiser Study Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3215 patients were screened for enrollment, and 405 did not proceed in the study. Participants were randomized in a 2:2:1 ratio.
Groups:
- Mucinex 2400 mg/Day: The study is designed to meet regulatory requirement outside the US. The dosing regimen and assessments timepoints were dictated by IR GGE and do not match approved Mucinex labeling. Participants were instructed to take 2 Mucinex (600-mg) tablets and 1 placebo tablet matching the 200-mg IR guaifenesin tablet by mouth, every 12 hours for 7 days. To ensure complete blinding, on Hours 6 and 18, this treatment group took 2 matching Mucinex placebo tablets combined with 1 IR guaifenesin placebo tablet.
Period: Overall Study
Arm/Group | Mucinex 2400 mg/Day | Immediate-release Guaifenesin 800 mg/Day | Placebo
Started | 1123 | 1124 | 563
Safety Population | 1122 | 1122 | 561
Modified Intent to Treat Population | 1106 | 1109 | 556
Completed | 1084 | 1086 | 547
Not Completed | 39 | 38 | 16
Not completed — Adverse Event | 5 | 2 | 2
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Lost to Follow-up | 17 | 15 | 9
Not completed — Protocol Violation | 3 | 2 | 2
Not completed — Withdrawal by Subject | 6 | 11 | 3
Not completed — Physician Decision | 5 | 6 | 0
Not completed — Sponsor decision | 0 | 1 | 0
Not completed — Assigned but never dosed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Based on the Safety population, defined as all patients who received at least one dose of the study medication, excluding patients who later return all the dispensed study medication to the site unused.
Groups:
- Mucinex 2400 mg/Day: The study is designed to meet regulatory requirement outside the US. The dosing regimen and assessments timepoints were dictated by IR GGE and do not match approved Mucinex labeling. Participants were instructed to take 2 Mucinex 600-mg tablets and 1 placebo tablet matching the 200 mg IR guaifenesin tablet by mouth, every 12 hours for 7 days. To ensure complete blinding, on Hours 6 and 18, this treatment group took 2 matching Mucinex placebo tablets combined with 1 IR guaifenesin placebo tablet.
- Total: Total of all reporting groups
Arm/Group | Mucinex 2400 mg/Day | Immediate-release Guaifenesin 800 mg/Day | Placebo | Total
Number analyzed (Participants) | 1122 | 1122 | 561 | 2805
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.81) | 36.8 (13.81) | 37.9 (14.09) | 37.2 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 670 | 668 | 333 | 1671
  Male | 452 | 454 | 228 | 1134
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 7 | 2 | 10
  Asian | 31 | 25 | 13 | 69
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 3 | 10
  Black or African American | 382 | 419 | 200 | 1001
  White | 686 | 656 | 327 | 1669
  Other | 18 | 12 | 16 | 46

OUTCOME MEASURES:

1. Primary Outcome: Summary Scores on the SUM8 Daily Cough and Phlegm Diary Card On the Morning of Day 4
Description: Participants completed diary cards twice a day that asked questions about their cough and phlegm status. The Daily Cough and Phlegm Diary Card consisted of eleven questions, eight core questions plus three questions that were answered dependent upon the response to core questions. The SUM8 consisted of the sum of the answers to the eight core questions. Each question was answered on a scale of 0-4, with 4 representing the greatest severity of symptoms. The SUM8 thus had a scale range of 0-32 with 0 representing best possible symptoms, and 32 representing greatest severity of symptoms.
Time Frame: Day 4
Population: Modified Intent-To-Treat (i.e., all randomized and treated subjects who had a baseline and at least 1 post-baseline set of assessments). Only participants who completed Daily Cough and Phlegm Diary Cards on the morning of Day 4 are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mucinex 2400 mg/Day | Immediate-release Guaifenesin 800 mg/Day | Placebo
Number analyzed (Participants) | 1064 | 1081 | 542
units on a scale | 12.96 (6.226) | 12.87 (6.078) | 12.71 (5.828)

2. Primary Outcome: Summary Scores on the SUM8 Daily Cough and Phlegm Diary Card On the Morning of Day 5
Description: as for outcome 1
Time Frame: Day 5
Population: Modified Intent-to-Treat(i.e., all randomized and treated subjects who had a baseline and at least 1 post-baseline set of assessments). Only participants who completed Daily Cough and Phlegm Diary Cards on the morning of Day 5 are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mucinex 2400 mg/Day | Immediate-release Guaifenesin 800 mg/Day | Placebo
Number analyzed (Participants) | 1065 | 1060 | 537
units on a scale | 10.92 (6.448) | 10.80 (6.261) | 11.05 (5.900)

ADVERSE EVENTS:
Time Frame: Treatment-emergent timeframe: Day 1 to Day 7
Description: The safety population included all patients who received the study medication, excluding patients who later returned all the dispensed study medication to the site.
Arm/Group | Mucinex 2400 mg/Day | Immediate-release Guaifenesin 800 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1122 | 0/1122 | 1/561
Other Adverse Events (participants affected / at risk) | 84/1122 | 85/1122 | 41/561
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mucinex 2400 mg/Day (N=1122) | Immediate-release Guaifenesin 800 mg/Day (N=1122) | Placebo (N=561)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mucinex 2400 mg/Day (N=1122) | Immediate-release Guaifenesin 800 mg/Day (N=1122) | Placebo (N=561)
Diarrhoea (Gastrointestinal disorders) | 21 | 17 | 9
Nausea (Gastrointestinal disorders) | 18 | 19 | 6
Vomiting (Gastrointestinal disorders) | 7 | 3 | 4
Pyrexia (General disorders) | 2 | 5 | 3
Dizziness (Nervous system disorders) | 10 | 8 | 3
Headache (Nervous system disorders) | 22 | 27 | 11
Somnolence (Nervous system disorders) | 4 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less